CLINICAL TRIAL: NCT03887910
Title: Northwell Health Visits: A Family Connects Pilot Implementation at Northwell Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 18-0328
Record Dates: First submitted 2019-03-06; First posted 2019-03-25 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Unspecified Child Maltreatment, Suspected; Unspecified Child Maltreatment, Confirmed; Postpartum Depression
Keywords: Postpartum Nurse Home Visitation; Infant Emergency Medical Care Presentations; Mother Emergency Medical Care Presentations; Parent-Child Relationship Quality; Family Connections to Community Resources; Child Development and Milestone Achievement; Maternal Mental Health; Child Abuse; Child Neglect; Child Well-Care Compliance; Mother Well-Care Compliance
MeSH Terms: conditions — Depression, Postpartum | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Principal Investigator, Co-Investigator and Outcomes Assessors are Masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Intervention (Experimental): Northwell Health Visits postnatal Nurse Practitioner home visitation program and referrals and developmental toys.
  Interventions: Other: Enhanced Intervention
- Intervention (Experimental): Northwell Health Visits postnatal Nurse Practitioner home visitation program and developmental screening and parent guides only.
  Interventions: Other: Intervention
- Control (No Intervention): Usual care with developmental toys.

INTERVENTIONS:
Other: Enhanced Intervention — Participants randomized to the Enhanced Intervention group will receive the Family Connects program, an evidence- based structure that begins at the birthing hospital stay, followed by 1 to 3 nurse home visits between 4 to 12 weeks of infant age, a follow-up contact one month later and a discharge home visit six months later and a final follow-up contact one month after that. During the home visits, the nurse engages with the mother and completes a holistic health and psychosocial assessment, during which the unique risks and family needs across 12 family domains are evaluated and addressed with either referrals with matched community resources or thorough education. In addition, they will be given a set of six developmental toys.
  Other Names: Family Connects Plus Developmental Toys
  Arms: Enhanced Intervention
Other: Intervention — Participants randomized to the Intervention group will receive the Family Connects program, an evidence- based structure that begins at the birthing hospital stay, followed by 1 to 3 nurse home visits between 4 to 12 weeks of infant age, a follow-up contact one month later and a discharge home visit six months later and a final follow-up contact one month after that. During the home visits, the nurse engages with the mother and completes a holistic health and psychosocial assessment, during which the unique risks and family needs across 12 family domains are evaluated. For each screened domain, the nurse is able to systematically address them, which may result in an immediate intervention; either referrals with matched community resources or thorough education.
  Other Names: Family Connects
  Arms: Intervention

SUMMARY:
Northwell Health Visits (NHV) is a three year pilot replication of the evidence-based model, Family Connects, which is a brief universal Nurse Practitioner home visiting program for new mothers and their infants. We seek to compare outcomes among mothers and infants enrolled in the NHV enhanced intervention arm, those enrolled in the NHV screening-only arm, and those in the control arm. NHV will follow a three- armed randomized control trial design.

DETAILED DESCRIPTION:
Northwell Health Visits (NHV) is based on Family Connects (formerly Durham Connects), which is a short-term, universal, inexpensive postnatal nurse home visiting program designed to provide brief parenting intervention and to connect families with community resources based on individualized assessments of family needs. The intervention was found to reduce the number of infant emergency medical care episodes and rates of anxiety in mothers, as well as increase community connection, positive parenting behaviors, participation in higher quality out-of-home child care when implemented in Durham, so we are looking to replicate these outcomes. We are adapting the model to serve the local population that is served by Northwell Health - Katz Women's Hospital at Long Island Jewish (LIJ) Medical Center, to see if increasing services in and around discharge is more useful for mothers and infants, and improves outcomes for infants. The focus is of early intervention (education and support by Nurse Practitioner), and connection to community agencies, in order to: reduce healthcare costs, decrease the rate of mothers and infants Potentially Preventable Emergency Room Visits (PPVs), adhere to well-baby care and mother's postpartum care schedules, improve family functioning, strengthen family partnerships and well-being, reduce necessary reports to child protective services, improve mental and physical health outcomes of mothers and infants within the first six months of life.

ELIGIBILITY:
Inclusion Criteria:

* Infant Born at Katz Women's Hospital at Long Island Jewish (LIJ) Medical Center
* Mother Age 18 years or older
* Mother who has delivered a single live born normal infant, vaginally or by cesarean section
* Mother Primary Language Spoken is English

Exclusion Criteria:

* Loss of Pregnancy
* Fetal demise
* No health insurance
* Infant in neonatal intensive care unit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Child Emergency Room Presentation Rates | Program enrollment until 24 months of Child Age.
  As reported in hospital administrative records and reported by parent.
Mother Emergency Room Presentation Rates | Program enrollment until 24 months postnatal.
  As reported in hospital administrative records and self report.
Child Hospital Admissions | Program enrollment until 24 months postnatal.
  As reported in hospital administrative records and reported by parent.
Mother Hospital Admissions | Program enrollment until 24 months postnatal.
  As reported in hospital administrative records and self report.

SECONDARY OUTCOMES:
Mother Postnatal Well-Care Compliance Rates | Program enrollment until 24 months postnatal.
  Rates of mother compliance with postnatal well-care, self reported and found on hospital records.
Child Postnatal Well-Care Compliance Rates | Program enrollment until 24 months postnatal.
  Rates of infant compliance with postnatal well-care health checks as reported by mother and found on hospital records.
Mother Mental Health - Anxiety Rates | Program enrollment until 24 months postnatal.
  Rates of postpartum anxiety symptoms as reported by mother. Assessed with General Anxiety Disorder-7 (GAD-7).
  Generalized Anxiety Disorder 7-Item (GAD-7) Scale Over the last 2 weeks, how often have you been bothered by the following problems?
  1. Feeling nervous, anxious, or on edge
  2. Not being able to stop or control worrying
  3. Worrying too much about different things
  4. Trouble relaxing
  5. Being so restless that it's hard to sit still
  6. Becoming easily annoyed or irritable
  7. Feeling afraid as if something awful might happen
  Score each with the following options:
  Not at all (0) Several days (1) More than half the days (2) Nearly every day (3) Scoring Criteria: Total score (adding all the numbers) provides a possible score from 0-21.
  GAD-7 Total Score Symptom Range 0-4 Minimal Anxiety 5-9 Mild Anxiety 10-14 Moderate Anxiety 15-21 Severe Anxiety
Mother Mental Health - Depression Rates | Program enrollment until 24 months postnatal.
  Rates of postpartum depression symptoms as reported by mother. Assessed with Edinburgh Postnatal Depression Scale (EPDS).
  SCORING QUESTIONS 1, 2, & 4 (without an *) Are scored 0, 1, 2 or 3 with top box scored as 0 and the bottom box scored as 3.
  QUESTIONS 3, 510 (marked with an *) Are reverse scored, with the top box scored as a 3 and the bottom box scored as 0.
  Maximum score: 30 Possible Depression: 10 or greater Always look at item 10 (suicidal thoughts)
Family Connections to Community Services/Resources | Program enrollment until 7 months postnatal.
  Rates of family connections to community resources and services as reported by the mother.
Mother parenting behaviors | Program enrollment until 24 months postnatal.
  Rates of mother positive and negative parenting behaviors as reported by mother.
Mother alcohol and other drug abuse | Program enrollment until 24 months postnatal.
  Rates of mother alcohol and other drug abuse as reported by mother and assessed using CAGE-AID screening tool.
  The CAGE questionnaire is used to test for alcohol abuse and dependence in adults. The CAGEAID version of the tool has been adapted to include drug use. Item responses on the CAGE and CAGE-AID are scored 0 or 1, with a higher score indicating alcohol or drug use problems. Each affirmative response earns one point. One point indicates a possible problem. Two points indicate a probable problem. 2/4 or greater = positive CAGE, further evaluation is indicated.
Family Violence | Program enrollment until 24 months postnatal.
  Rates of family violence as assessed using the Conflict Tactics Scale (CTS). Instructions: Please check the answer that best describes your relationship with your partner in the past year? The CTS is scored by adding the midpoints for the response categories chosen by the participant. The midpoints are the same as the response category numbers for Categories 0, 1, and 2. For Category 3 (3-5 times) the midpoint is 4, for Category 4 (6- or more times) it is 8.
  A score of 0 is negative for family violence,higher scores are indicative of greater physical abuse

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health, Manhasset, New York, United States

REFERENCES:
- [Derived] Yonemoto N, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2021 Jul 21;7(7):CD009326. doi: 10.1002/14651858.CD009326.pub4. PMID 34286512